CLINICAL TRIAL: NCT05309083
Title: Moving Mindfully: A MBSR-Centered Approach to Freezing in Parkinson Disease
Brief Title: Moving Mindfully for Freezing in Parkinsons
Acronym: MMR34
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Gammon M Earhart, Professor, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202012021
Record Dates: First submitted 2022-03-16; First posted 2022-04-04 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease; Freezing of Gait
Keywords: Mindfulness
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: In Aim 2, participants will receive the mindfulness intervention as part of the open pilot.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Based Walking Therapy (MBWT) (Experimental): Participants will participate in MBWT.
  Interventions: Behavioral: Mindfulness Based Walking Therapy (MBWT)

INTERVENTIONS:
Behavioral: Mindfulness Based Walking Therapy (MBWT) — MBWT will be a modified form of the typical Mindfulness Based Stress Reduction (MBSR) program that incorporates more walking meditations and is acceptable for people with Parkinson disease and freezing of gait.

SUMMARY:
The investigators will modify and evaluate the feasibility of a mindfulness intervention among people living with Parkinson disease (PD) and freezing of gait (FOG). FOG is a severe motor disturbance that prevents people from stepping normally and is associated with anxiety, frustration, sedentary behaviors, poorer quality of life, and falls. Mindfulness-Based Stress Reduction (MBSR) is an evidence-based practice that creates a culture to reduce stress and anxiety by increasing conscious awareness and self-compassion. In this study, the investigators will develop a mindfulness-based walking intervention to address both mental health and mobility challenges that constitute FOG. This R34 feasibility study includes three aims to permit the development of a mind and body approach for FOG among people living with PD.

DETAILED DESCRIPTION:
Aim 1: Create a Mindfulness-Based Walking Therapy (MBWT) program by modifying the MBSR standard protocol based upon feedback from an advisory group. An advisory group consisting of physical therapists, mindfulness instructors, research team members, 3-5 people with PD+FOG and care partners will modify the standard MBSR program over a twelve-week period to make it acceptable and feasible for people with PD+FOG and shift the focus from sitting, standing, or lying meditations to walking mediations.

Aim 2: Refine and standardize the MBWT protocol to ensure feasibility and acceptability through open pilot testing. Twelve participants with PD+FOG will participate in an open pilot of the MBWT program. The MBWT program will then be modified based on participant feedback to produce a standardized MBWT to use in Aim 3. Feasibility elements include meeting benchmarks for: 1) recruitment and randomization; 2) retention and satisfaction; 3) delivery of the intervention; 4) participant adherence using technology; 5) evaluating clarity and burden of outcome assessments; and 6) monitoring adverse events.

Aim 3: Conduct pilot randomized clinical trial to evaluate feasibility and acceptability of the standardized MBWT program. Using the standardized MBWT protocol produced from Aim 2, the investigators will randomize 24 people with PD+FOG to MBWT or usual care (i.e., medical management and FOG education), examining feasibility elements listed in Aim 2. The investigators will also conduct follow-up evaluations to monitor burden and continued usage of mindfulness. Aim 3 is under NCT05923229.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed by a neurologist with idiopathic Parkinson disease;
* age 55 and older;
* a score on the Hoehn & Yahr (H&Y) scale between I-IV;
* history of freezing of gait;
* able to provide informed consent;
* experience fear or worry in relation to their freezing of gait;
* able to walk independently with or without an assistive device for at least five minutes; and
* stable medication regimen for two months prior to enrollment.

Exclusion Criteria:

* have evidence of dementia (Montreal Cognitive Assessment (MOCA) < 18) to ensure understanding of materials;
* are under consideration for deep brain stimulation surgery within the next six months;
* neurologic condition other than PD;
* inability to cooperate with the protocol;
* language, visual, or hearing barriers to participation; or
* history of orthopedic or other medical problems that limit ability to participate safely in the intervention.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gammon Earhart, PT, PhD, Principal Investigator — Washington University School of Medicine; Kerri Rawson, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine Program in Physical Therapy, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness Based Walking Therapy (MBWT)
Started | 9
Completed | 7
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- MBWT: Mindfulness-Based Walking Therapy Program
Arm/Group | MBWT
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.44 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
New Freezing of Gait Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The New Freezing of Gait Questionnaire quantifies severity of freezing of gait with a total range of 0 to 28. Higher scores indicate more severe freezing of gait.
  units on a scale | 16.78 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Recruitment of Sample: Number of Participants Recruited
Description: The investigators will count the number of participants recruited to determine if the feasibility objective of recruitment is met. The investigators benchmark for recruitment is defined as recruiting a target sample of 12 participants.
Time Frame: 14 weeks
Population: Twelve participants were recruited and signed a consent form. Three participants did not pass in-person screening resulting in nine participants who started the intervention.
Measure: Count of Participants; unit: Participants
Groups:
- MBWT: Mindfulness-Based Walking Therapy
Arm/Group | MBWT
Number analyzed (Participants) | 12
Participants | 12

2. Primary Outcome: Attendance of Participants: Average Percentage of Participants at Each Session
Description: The investigators will count the number of participants at each session and report the average percentage of participants that attended each session over the course of the study to determine if the feasibility objective of attendance is met. The investigators benchmark for attendance is defined as at least 80% of participants attending each session.
Time Frame: 14 weeks
Population: 7 participants completed the 14 week program, 2 participants withdrew after class 5
Measure: Mean (Full Range); unit: percentage of participants
Arm/Group | MBWT
Number analyzed (Participants) | 9
percentage of participants | 79.82 [55.56 to 100]

3. Primary Outcome: Retention of Participants: Average Percentage of Sessions Each Participant Completes
Description: The investigators will count the number of sessions each participant attends and report the number of classes each participant attended on average to determine if the feasibility objective of retention is met. The investigators benchmark for retention is defined as participants attending 80% of the sessions.
Time Frame: 14 weeks
Population: 7 participants who completed the 14 week program and 2 participants who withdrew after class 5
Measure: Mean (Full Range); unit: percentage of classes attended
Arm/Group | MBWT
Number analyzed (Participants) | 9
percentage of classes attended | 78.25 [60 to 100]

4. Primary Outcome: Adherence: Average Percentage of Hours Participants Practiced Mindfulness at Home
Description: The investigators will ask participants to track the number of hours spent practicing mindfulness at home to determine if the feasibility objective of adherence is met. The investigators benchmark for adherence is defined as participants completing 70% of daily home assignment hours.
Time Frame: 14 weeks
Population: Only five participants regularly reported home assignment hours.
Measure: Mean (Full Range); unit: percentage of home assignment hours
Arm/Group | MBWT
Number analyzed (Participants) | 5
percentage of home assignment hours | 147.84 [23 to 325]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during baseline evaluations (1-4 weeks prior), the 14 week intervention, post evaluations (1-4 weeks post intervention) and follow-up evaluations (12-16 weeks after post); on average 38 weeks.
Arm/Group | MBWT
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBWT (N=9)
Fall (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT05309083/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT05309083/ICF_001.pdf